CLINICAL TRIAL: NCT07284225
Title: A Randomized Controlled Study on the Acute Effects of a Single Dose of Nicotinamide Riboside on Sleep Structure in Healthy Adults
Brief Title: Acute Effects of Nicotinamide Riboside on Polysomnography-Measured Sleep Structure in Healthy Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2025287
Record Dates: First submitted 2025-11-30; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotinamide Riboside (NR) Group (Experimental): Participants randomized to this arm will receive a single oral dose of 600 mg NR approximately one hour before their second overnight PSG assessment.
  Interventions: Dietary Supplement: Nicotinamide Riboside (NR)
- Placebo Group (Placebo Comparator): Participants randomized to this arm will receive a matching placebo capsule approximately one hour before their second overnight PSG assessment. The placebo is identical in appearance to the NR capsule and contains inert ingredients without active pharmacological effects.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside (NR) — A single oral dose of 600 mg NR, an NAD+ precursor compound, provided in capsule form. The dose and timing are standardized for all participants.
  Arms: Nicotinamide Riboside (NR) Group
Other: Placebo — The placebo capsule is visually identical to the NR capsule but contains inert excipients without active pharmacological components.
  Arms: Placebo Group

SUMMARY:
This study aims to evaluate whether a single oral dose of nicotinamide riboside (NR), a precursor of nicotinamide adenine dinucleotide (NAD+), has acute effects on sleep in healthy adults who report mild sleep difficulties. NR is widely used as a nutritional supplement and is known to increase cellular NAD+ levels, which may influence physiological processes linked to sleep-wake regulation.

In this randomized, double-blind, placebo-controlled study, 20 healthy adults will complete two overnight sleep assessments using polysomnography (PSG), the gold-standard sleep monitoring method. After a baseline night of sleep recording, participants will receive either NR or a placebo before bedtime on the second night. Researchers will compare sleep duration and sleep structure before and after the intervention to determine whether NR has an acute effect on objective sleep quality.

The study will also evaluate safety and collect participants' subjective sleep impressions. Findings may help clarify whether NR, a widely used nutritional supplement, has measurable short-term effects on human sleep.

DETAILED DESCRIPTION:
Sleep quality is a major component of overall health, yet many adults experience mild but persistent sleep difficulties. Nicotinamide riboside (NR) is a naturally occurring precursor of NAD+, a key coenzyme involved in cellular energy metabolism and circadian regulation. Preclinical studies suggest that NR may influence neural pathways related to sleep-wake control, but its short-term, objective effects on human sleep architecture have not been well established.

This study is designed to explore the acute impact of NR on objectively measured sleep in healthy adults with mild subjective sleep complaints. It uses a randomized, double-blind, placebo-controlled design to minimize bias. All participants will spend two consecutive nights in a controlled sleep laboratory. The first night serves as a baseline assessment of natural sleep. On the second night, individuals will receive a single 600 mg dose of NR or a matched placebo one hour before bedtime.

Polysomnography (PSG) will be used to evaluate total sleep time, sleep stages, sleep efficiency, sleep latency, and wakefulness during the night. Subjective sleep quality will be assessed with validated questionnaires administered the morning after each sleep recording. Safety will be monitored throughout the study period and through a follow-up contact after discharge.This exploratory early-phase study aims to generate objective human data regarding the feasibility, safety, and potential sleep-modulating effects of NR.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females aged 18 to 60 years inclusive;
* Screening using the Pittsburgh Sleep Quality Index (PSQI) scale with a total score between 5 and 10, indicating mild subjective sleep disturbance;
* Voluntarily participate in this study and sign a written informed consent form;
* Able to understand the study procedures and willing to comply with all laboratory regulations.

Exclusion Criteria:

* History of any serious neurological, cardiovascular, respiratory, hepatic, renal, hematological, or psychiatric disorders;
* Medically diagnosed sleep disorders (e.g., insomnia, sleep apnea syndrome, restless legs syndrome);
* Regular use within the past month of any medication or supplement that may affect sleep (e.g., sedatives, antidepressants, antihistamines, melatonin);
* Known allergy to nicotinamide riboside (NR) or any component of the study product;
* History of chronic smoking, heavy alcohol consumption (exceeding weekly recommended intake), or substance abuse;
* Participation in any other interventional clinical studies within one month prior to study initiation, or exposure to circadian rhythm-disrupting factors such as trans-time zone travel or frequent night shifts;
* Pregnant women, breastfeeding women, or men of reproductive age with plans to conceive within the next month who are not using effective contraception.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Total Sleep Time (TST) | Measured during the baseline night (pre-intervention) and the experimental night (post-NR or placebo).
  Total amount of sleep obtained during the overnight PSG recording, measured in minutes.

SECONDARY OUTCOMES:
Sleep Latency | Measured during the baseline night (pre-intervention) and the experimental night (post-NR or placebo).
  Duration from lights-off to the first epoch of any sleep stage during PSG, measured in minutes.
Wake After Sleep Onset | Measured during the baseline night (pre-intervention) and the experimental night (post-NR or placebo).
  Total duration of wakefulness after initial sleep onset but before final awakening, measured in minutes via PSG.
Sleep Stage Distribution | Measured during the baseline night (pre-intervention) and the experimental night (post-NR or placebo)
  Minutes spent in N1, N2, N3, and REM sleep during overnight PSG, recorded as absolute minutes for each stage.
Leeds Sleep Evaluation Questionnaire | Morning of the day after the experimental night (approximately 8:00 AM).
  Self-reported subjective sleep quality assessed using the Leeds Sleep Evaluation Questionnaire (LSEQ). The outcome is reported as a total score ranging from 0 to 10, with higher scores indicating better perceived sleep quality and better condition upon awakening.

IPD SHARING:
Plan to Share IPD: No